CLINICAL TRIAL: NCT04330599
Title: Longitudinal Population-based Observational Study of COVID-19 in the UK Population
Acronym: COVIDENCE UK
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: King's College London (Other); London School of Hygiene and Tropical Medicine (Other); University of Edinburgh (Other); Swansea University (Other); Queen's University, Belfast (Other); Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: COVIDENCE UK
Record Dates: First submitted 2020-03-31; First posted 2020-04-01 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Eluates from dried blood spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVIDENCE UK is a population-based observational longitudinal study that has the following objectives:

1. To determine risk factors for incident COVID-19 and for adverse outcomes of COVID-19 in the UK population
2. To characterise the natural history of COVID-19 in the UK population
3. To evaluate the impact of COVID-19 on the physical and mental health of the UK population
4. To provide a resource from which to identify potential participants for future clinical trials, and to use data collected in COVIDENCE as comparison or control data for trial participants who have been randomised to receive one or more interventions.

ELIGIBILITY:
Inclusion Criteria:

* UK resident
* Age ≥16 years

Exclusion Criteria: none

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: UK residents aged 16 years or more
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of confirmed COVID-19 | 5 years

SECONDARY OUTCOMES:
Incidence of probable or suspected COVID-19 | 5 years
Incidence of COVID-19 requiring hospitalisation | 5 years
Incidence of COVID-19 requiring ventilatory support | 5 years
Incidence of fatal COVID-19 | 5 years
Symptom duration per COVID-19 episode | 5 years
Symptom severity per COVID-19 episode | 5 years
Incidence of seroconversion to SARS-CoV-2 | 5 years
Incidence of recurrent COVID-19 | 5 years
EQ-5D-3L health-related quality of life score | 5 years
Health care costs associated with incident COVID-19 | 5 years
Impact of the COVID-19 pandemic and the societal response on participants' financial status | 5 years
Incidence of COVID-19 on participant's physical health | 5 years
Impact of COVID-19 on participants' mental health | 5 years
Impact of COVID-19 on physical health of offspring born to participants during follow-up | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary University of London, London, County (optional), United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Vivaldi G, Talaei M, Blaikley J, Jackson C, Pfeffer PE, Shaheen SO, Martineau AR. Bidirectional relationship between sleep problems and long COVID: a longitudinal analysis of data from the COVIDENCE UK study. BMJ Open Respir Res. 2025 Jun 15;12(1):e002506. doi: 10.1136/bmjresp-2024-002506. PMID 40518292
- [Derived] Vivaldi G, Pfeffer PE, Talaei M, Basera TJ, Shaheen SO, Martineau AR. Long-term symptom profiles after COVID-19 vs other acute respiratory infections: an analysis of data from the COVIDENCE UK study. EClinicalMedicine. 2023 Oct 6;65:102251. doi: 10.1016/j.eclinm.2023.102251. eCollection 2023 Nov. PMID 38106559
- [Derived] Tydeman F, Pfeffer PE, Vivaldi G, Holt H, Talaei M, Jolliffe D, Davies G, Lyons RA, Griffiths C, Kee F, Sheikh A, Shaheen SO, Martineau AR. Rebound in asthma exacerbations following relaxation of COVID-19 restrictions: a longitudinal population-based study (COVIDENCE UK). Thorax. 2023 Aug;78(8):752-759. doi: 10.1136/thorax-2022-219591. Epub 2022 Nov 23. PMID 36423925
- [Derived] Williamson AE, Tydeman F, Miners A, Pyper K, Martineau AR. Short-term and long-term impacts of COVID-19 on economic vulnerability: a population-based longitudinal study (COVIDENCE UK). BMJ Open. 2022 Aug 23;12(8):e065083. doi: 10.1136/bmjopen-2022-065083. PMID 35998959
- [Derived] Holt H, Talaei M, Greenig M, Zenner D, Symons J, Relton C, Young KS, Davies MR, Thompson KN, Ashman J, Rajpoot SS, Kayyale AA, El Rifai S, Lloyd PJ, Jolliffe D, Timmis O, Finer S, Iliodromiti S, Miners A, Hopkinson NS, Alam B, Lloyd-Jones G, Dietrich T, Chapple I, Pfeffer PE, McCoy D, Davies G, Lyons RA, Griffiths C, Kee F, Sheikh A, Breen G, Shaheen SO, Martineau AR. Risk factors for developing COVID-19: a population-based longitudinal study (COVIDENCE UK). Thorax. 2022 Sep;77(9):900-912. doi: 10.1136/thoraxjnl-2021-217487. Epub 2021 Nov 30. PMID 34848555